CLINICAL TRIAL: NCT03760055
Title: Assessment of Visual Function With a Portable Brain-computer Interface
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: NGoggle (Industry)
Collaborators: Duke University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00100894; R42EY027651 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma; Age Related Macular Degeneration; Optic Neuropathy; Retinal Degeneration
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Optic Nerve Diseases; Retinal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Glaucoma and glaucoma suspects: Patients with at least two consecutive and reliable standard automated perimetry (SAP) examinations with either a pattern standard deviation (PSD) outside the 95% normal limits or a glaucoma hemifield test (GHT) result outside the 99% normal limits. Patients considered suspects for glaucoma must have an intraocular pressure (IOP) greater than 21 millimeters of mercury (mmHg) or suspicious appearance of the optic nerve head but with reliable normal visual fields, defined as a PSD within 95% confidence limits and a GHT result within normal limits.
  Interventions: Device: nGoggle
- Age-related macular degeneration: Patients will be considered as having AMD if one or more of the following are present on posterior biomicroscopy (fundoscopy), indirect ophthalmoscopy or Optical Coherence Tomography (OCT) exams:
  1. Presence of at least intermediate-size drusen (63µm or larger in diameter)
  2. Retinal pigment epithelium (RPE) abnormalities such as hypopigmentation or hyperpigmentation
  3. Reticular pseudodrusen (also called sub retinal drusenoid deposit)
  4. Presence of any of the following features: geographic atrophy of the RPE, choroidal neovascularization (exudative, wet), polypoidal choroidal vasculopathy, or retinal angiomatous proliferation.
  Interventions: Device: nGoggle
- Other eye diseases: Patients with other retinal degenerations such as retinitis pigmentosa or with other diseases affecting the visual pathways such as tumors, ischemic neuropathy or optic neuritis may also be included. Their diagnosis will be extracted from their clinical visits.
  Interventions: Device: nGoggle
- Healthy subjects: To be considered healthy, subjects have to have IOP < 22 mmHg with no history of elevated IOP and with at least two reliable normal visual fields, defined as a PSD within 95% confidence limits and a GHT result within normal limits.
  Interventions: Device: nGoggle

INTERVENTIONS:
Device: nGoggle — The nGoggle is a portable visual evoked potential system that uses an EEG to acquire visual evoked potentials in response to visual stimuli presented on a virtual reality goggle. The investigators will assess the ability of the nGoggle to detect visual field loss in patients with glaucoma, as well as to discriminate among the different stages of the disease, its repeatability and reliability for patient self-testing and patient satisfaction compared to standard automated perimetry (SAP), optical coherence tomography (OCT) metrics and Diopsys NOVA (Diopsys, Inc.). In addition, patients with other diseases affecting the visual system will also be tested in order to assess whether the nGoggle can differentiate glaucoma from them.
  Other Names: Portable brain-computer interface

SUMMARY:
1. The purpose of this study is to evaluate the nGoggle's accuracy and repeatability in detecting visual function loss. In addition, the ability to stage glaucomatous damage and investigate the relationship between nGoggle metrics and neural damage in glaucoma will also be evaluated.
2. Longitudinal study, including 200 patients with: glaucoma, suspected of having glaucoma, nonglaucomatous optic neuropathies, AMD, retinal degenerations, other diseases involving the visual pathways, besides healthy controls. Subjects will perform standard ophthalmological exams, and the following research tests: electroencephalogram, visual evoked potentials, and questionnaires.
3. Statistical analyses will be performed by the PI using the software Stata, MATLAB, and MPLUS. Risks are low, consisting of some discomfort, fatigue, dizziness or motion sickness.

DETAILED DESCRIPTION:
Background & Significance

Assessment of functional loss in glaucoma has been traditionally made with standard automated perimetry (SAP). Despite the significant progress achieved with the development of SAP, assessment of visual field loss still has significant drawbacks. SAP testing is limited by subjectivity of patient responses and high test-retest variability, frequently requiring many tests for effective detection of change over time. Moreover, as these tests are generally conducted in clinic-based settings, limited patient availability and health care resources often result in an insufficient number of tests acquired over time, with delayed diagnosis and detection of disease progression. The requirement for highly trained technicians, cost, complexity, and lack of portability of SAP also preclude its use for screening of visual field loss in underserved populations. Furthermore, current SAP testing as performed in clinical practice frequently results in delayed detection of progression, with potential late initiation/escalation of treatment and irreversible functional damage.

As a part of a funded Phase I project, the nGoggle (nGoggle Inc., San Diego, CA), the first device of its kind, allowed a portable and objective brain-based assessment of visual function deficits in glaucoma. The nGoggle integrates a wearable, wireless, no-prep EEG system and a head-mounted display (HMD) to allow users to routinely monitor electrical brain activities associated with visual field stimulation. A recent study comparing the diagnostic accuracies of an earlier version of the nGoggle and SAP in discriminating patients with glaucoma from healthy subjects found that the nGoggle performed at least as well, if not better than, SAP with the additional advantage of portability and objectivity.

The overall goal of this proposal is to test the nGoggle's accuracy and repeatability in detecting visual function loss. In addition, its ability to stage glaucomatous damage, by discriminating patients at different stages of the disease will be evaluated. Finally, the relationship between nGoggle metrics and neural damage in glaucoma as detected by other objective techniques such as optical coherence tomography will also be investigated. Patients with other diseases affecting the visual system will also be included in order to assess whether the nGoggle can differentiate glaucoma from them.

Study Design & Procedures

This will be a longitudinal study in which patients will be examined approximately biannually. The following patients will be recruited:

1. Glaucoma;
2. Suspicion of having glaucoma;
3. Non-glaucomatous optic neuropathies;
4. Age-related macular degeneration (AMD);
5. Retinal degenerations;
6. Other diseases involving the visual pathways such as optic neuritis, tumors or ischemic neuropathy.
7. Healthy subjects

General evaluation:

As part of the study all participants will undergo the following general evaluation:

1. Review of medical history;
2. Comprehensive ophthalmologic examination
3. Questionnaires: a. Cognitive function using the Montreal Cognitive Assessment (MoCA); b. A short structured interview to obtain vision-related quality of life information using the National Eye Institute 25-Item Visual Functioning Questionnaire (NEI VFQ-25); c. A questionnaire to assess patient's satisfaction with the nGoggle testing, including easiness of placement, comfort, and user-interface.
4. Electroencephalogram (EEG) and Visual Evoked Potentials (VEP): Visual evoked potentials (VEP) will be evaluated with Diopsys NOVA (Diopsys, Inc.), which is a well-established conventional multifocal VEP device to assess brain functioning following visual stimuli from a computer screen. Subjects will also be monitored with an EEG system integrated with a head-mounted display (nGoggle, Inc.). The nGoggle is a portable visual evoked potential system that uses an EEG to acquire visual evoked potentials in response to visual stimuli presented on a virtual reality goggle.

Risk/Benefit Assessment

Risks:

Risks from participating in the study are very low. The primary risks for all participants are some discomforts, which are similar to those encountered in any complete eye examination. Participants will undergo non-invasive procedures used for diagnostic purposes that are used in standard clinical care. Eventually, it will be necessary to use numbing or dilating drops for fundus examination, as is done in standard clinical care. Some risks of those drops include: dry eye, mild headache, blurred vision, drowsiness, burning eyes, tearing, light sensitivity, redness, and allergy reactions. The only non-FDA approved device used in this study is the nGoggle (nGoggle Inc.), which is an investigational diagnostic device qualified as a non-significant risk device. The subject may experience mild discomfort due to drying of the eye during the study. Should a patient note drying, a drop of artificial tears will be placed over the eye by the study key personnel. In very rare cases, artificial eye tear drops may cause irritation or allergy. There are no known risks associated with the EEG test other than discomfort and fatigue. Subjects might become bored, fatigued or distressed while participating. To minimize these potential effects, the tasks will be kept short and subjects will be instructed that they may request to interrupt the test anytime. All assessments, software, instruments that are not FDA approved will be used as tools to assess disability and device efficacy, and will not be used as a diagnostic procedure without confirmation of the diagnosis by another, medically established diagnostic product or procedure. There is, however, the potential risk of loss of confidentiality. Every effort will be made to keep the information confidential; however, this cannot be guaranteed. Some of the questions that will be asked as part of this study may make the patients feel uncomfortable. Patients may refuse to answer any of the questions and may take a break at any time during the study. Patient may stop their participation in this study at any time.

Unknown/unforeseeable risks

In addition to the risks and discomforts listed here, there may be other risks that are currently not known. Subjects will be informed if any other potential risk becomes known through the duration of the study. Also, the risks and discomforts may occur more often or be more severe than have been seen before and written in this form.

Benefits:

Subjects will be referred from the Duke Eye Center care providers after a comprehensive clinical eye examination from a routine visit. If the last clinical eye examination is not within 6 months of the study visit, the participant will be examined by the PI, with no additional cost to the patient.

Participants will also undergo tests that will allow the validation and development of a transformative device for diagnosing and monitoring ocular diseases, and could be suited for home-based testing of visual function in the future, which could benefit patients with eye diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 90 years old;
2. Both males and females will be included.
3. Be able and willing to provide signed informed consent and follow study instructions

Exclusion Criteria:

1. Subjects will be excluded if they present with any systemic or ocular conditions that in the opinion of the Principal Investigator may prevent them from completing the tests (e.g. history of seizures or other coexistent ocular pathologies).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The following patients will be recruited from Dr. Tseng's clinic by verbal communication. Staff members at the Duke Eye Center will also be invited to recommend potential participants for the study, in conformance with the Duke Human Subjects Committee Guidelines.
  1. Glaucoma;
  2. Suspicion of having glaucoma;
  3. Non-glaucomatous optic neuropathies;
  4. Age-related macular degeneration (AMD);
  5. Retinal degenerations;
  6. Other diseases involving the visual pathways such as optic neuritis, tumors or ischemic neuropathy.
  7. Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Device accuracy to detect visual field loss | from date of enrollment and every 6 months, up to 5 years
  Comparison of diagnostic accuracies will be performed by analyzing areas under the receiver operating characteristic (ROC) curves for each nGoggle and SAP metric by assessment of partial areas under the ROC curves (targeting high specificity>90% region), sensitivities at matched specificities and diagnostic likelihood ratios (LRs). The investigators will also evaluate the correlation between nGoggle multifocal steady-state visual evoked potentials (mfSSVEP) metrics and SAP parameters throughout the disease spectrum.
Device accuracy to detect structural neural loss | from date of enrollment and every 6 months, up to 5 years
  Comparison of diagnostic accuracies will be performed by analyzing areas under the receiver operating characteristic (ROC) curves for each nGoggle and OCT parameters, as well as by assessment of partial areas under the ROC curves (targeting high specificity>90% region), sensitivities at matched specificities and diagnostic likelihood ratios (LRs). The investigators will also evaluate the correlation between nGoggle mfSSVEP metrics and SDOCT parameters throughout the disease spectrum. SDOCT testing will be performed with Spectralis OCT (Heidelberg Engineering, Germany). SDOCT parameters to be investigated will include retinal nerve fiber layer (RNFL) thickness, minimum rim width (MRW) and macular thickness.
Device accuracy to detect objective functional loss | from date of enrollment and every 6 months, up to 5 years
  Comparison of diagnostic accuracies will be performed by analyzing areas under the receiver operating characteristic (ROC) curves for each nGoggle and Diopsys NOVA parameters, as well as by assessment of partial areas under the ROC curves (targeting high specificity>90% region), sensitivities at matched specificities and diagnostic likelihood ratios (LRs). The investigators will also evaluate the correlation between nGoggle mfSSVEP metrics and those parameters throughout the disease spectrum. SDOCT testing will be performed with Spectralis OCT (Heidelberg Engineering, Germany). SDOCT parameters to be investigated will include retinal nerve fiber layer (RNFL) thickness, minimum rim width (MRW) and macular thickness.
Assessment of repeatability | 6 weeks
  Assessment of repeatability of the device parameters will be evaluated through intra-class correlation coefficient (ICC). A subgroup of subjects will undergo 5 visits over a short period of time (6 weeks). A sample size of 35 subjects will provide a width of 0.1 for the 95% for ICC, allowing assessment of repeatability of the devices parameters.

SECONDARY OUTCOMES:
Patients' satisfaction | from date of enrollment and every 6 months, up to 5 years
  The investigators will obtain a survey regarding patients' satisfaction with testing, including easiness of placement, comfort, and user-interface.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Tseng, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.